CLINICAL TRIAL: NCT02084706
Title: Needle-Free Injection of Lidocaine for Local Anesthesia Prior to Trigger Digit Injection
Acronym: J-tip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Philip Blazar, MD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2013P002370
Record Dates: First submitted 2014-03-05; First posted 2014-03-12 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Triamcinolone; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triamcinolone (20 g) and 2% Lidocaine injection over A1 pulley (Active Comparator): Group one subjects will receive an injection of 0.5mL (20 g) of Triamcinolone and 0.5 mL of 2% Lidocaine over the A1 pulley.
  Interventions: Procedure: Triamcinolone (20 g) and 2% Lidocaine injection over the A1 pulley; Drug: 2% Lidocaine; Drug: Triamcinolone (20 g)
- J-tip lidocaine administration, then steroid injection (Experimental): Group two subjects will receive a needle free "J-tip" administration of 0.5mL of 2% lidocaine prior (2-10 minutes) to needle injection of 0.5mL of Triamcinolone (20 g) over the A1 pulley.
  Interventions: Drug: 2% Lidocaine; Drug: Triamcinolone (20 g); Procedure: J-tip lidocaine administration; Procedure: Triamcinolone (20 g) Injection over the A1 pulley.

INTERVENTIONS:
Procedure: Triamcinolone (20 g) and 2% Lidocaine injection over the A1 pulley
  Arms: Triamcinolone (20 g) and 2% Lidocaine injection over A1 pulley
Drug: 2% Lidocaine
Drug: Triamcinolone (20 g)
Procedure: J-tip lidocaine administration
  Arms: J-tip lidocaine administration, then steroid injection
Procedure: Triamcinolone (20 g) Injection over the A1 pulley.
  Arms: J-tip lidocaine administration, then steroid injection

SUMMARY:
Jet-injection (J-tip) is a rapid, minimally invasive delivery system that can be used for the subdermal injection of lidocaine solution for anesthetic purposes. The device has been found effective in pain reduction during IV catheterization in adults and children and lumbar puncture in children when compared to placebo saline-jet injection. [1-4].

We believe that administering local anesthetic via J-tip prior to triamcinolone(40 mg/ml) injection could mitigate pain that occurs during and immediately following injection while preserving the post-injection pain relief of anesthetic injection. Furthermore, pre-placement of the jet-injected local anesthetic may obviate the need for the inclusion of local anesthetic into the triamcinolone injection. This would decrease the amount of fluid injected, which could have positive pain modulation by decreased tissue disruption.

Objective: To evaluate the effectiveness of needle free jet injection (J-tip) administration of 2% lidocaine in reduction of the pain experienced during trigger digit 40 mg/ml triamcinolone injection.

Hypothesis: Needle free jet injection (J-tip) administration of 2% lidocaine will prove an equal or superior means of pain reduction when compared to 2% lidocaine injection in the setting of trigger digit triamcinolone injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the Hand Clinic at Brigham and Women's Hospital or Brigham and Women's Faulkner Hospital, are 18 years of age or older and are indicated for a trigger digit steroid injection will be eligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Blazar, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lysakowski C, Dumont L, Tramer MR, Tassonyi E. A needle-free jet-injection system with lidocaine for peripheral intravenous cannula insertion: a randomized controlled trial with cost-effectiveness analysis. Anesth Analg. 2003 Jan;96(1):215-9, table of contents. doi: 10.1097/00000539-200301000-00044. PMID 12505955
- [Background] Ferayorni A, Yniguez R, Bryson M, Bulloch B. Needle-free jet injection of lidocaine for local anesthesia during lumbar puncture: a randomized controlled trial. Pediatr Emerg Care. 2012 Jul;28(7):687-90. doi: 10.1097/PEC.0b013e31825d210b. PMID 22743744
- [Background] Jimenez N, Bradford H, Seidel KD, Sousa M, Lynn AM. A comparison of a needle-free injection system for local anesthesia versus EMLA for intravenous catheter insertion in the pediatric patient. Anesth Analg. 2006 Feb;102(2):411-4. doi: 10.1213/01.ane.0000194293.10549.62. PMID 16428534
- [Background] Spanos S, Booth R, Koenig H, Sikes K, Gracely E, Kim IK. Jet Injection of 1% buffered lidocaine versus topical ELA-Max for anesthesia before peripheral intravenous catheterization in children: a randomized controlled trial. Pediatr Emerg Care. 2008 Aug;24(8):511-5. doi: 10.1097/PEC.0b013e31816a8d5b. PMID 18645542
- [Background] Kolind-Sorensen V. Treatment of trigger fingers. Acta Orthop Scand. 1970;41(4):428-32. doi: 10.3109/17453677008991530. No abstract available. PMID 5537268
- [Background] Lapidus PW, Guidotti FP. Stenosing tenovaginitis of the wrist and fingers. Clin Orthop Relat Res. 1972 Mar-Apr;83:87-90. doi: 10.1097/00003086-197203000-00015. No abstract available. PMID 5014835
- [Background] Rhoades CE, Gelberman RH, Manjarris JF. Stenosing tenosynovitis of the fingers and thumb. Results of a prospective trial of steroid injection and splinting. Clin Orthop Relat Res. 1984 Nov;(190):236-8. PMID 6488636
- [Background] Murphy D, Failla JM, Koniuch MP. Steroid versus placebo injection for trigger finger. J Hand Surg Am. 1995 Jul;20(4):628-31. doi: 10.1016/S0363-5023(05)80280-1. PMID 7594291

RESULTS

PARTICIPANT FLOW:
Groups:
- Triamcinolone (20 g) and 2% Lidocaine Injection Over A1 Pulley: Group one subjects will receive an injection of 0.5mL (20 g) of Triamcinolone and 0.5 mL of 2% Lidocaine over the A1 pulley.
  Triamcinolone (20 g) and 2% Lidocaine injection over the A1 pulley
  2% Lidocaine
  Triamcinolone (20 g)
- J-tip Lidocaine Administration, Then Steroid Injection: Group two subjects will receive a needle free "J-tip" administration of 0.5mL of 2% lidocaine prior (2-10 minutes) to needle injection of 0.5mL of Triamcinolone (20 g) over the A1 pulley.
  2% Lidocaine
  Triamcinolone (20 g)
  J-tip lidocaine administration
  Triamcinolone (20 g) Injection over the A1 pulley.
Period: Overall Study
Arm/Group | Triamcinolone (20 g) and 2% Lidocaine Injection Over A1 Pulley | J-tip Lidocaine Administration, Then Steroid Injection
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone (20 g) and 2% Lidocaine Injection Over A1 Pulley | J-tip Lidocaine Administration, Then Steroid Injection | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 27
  >=65 years | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (11.2) | 65.4 (10.3) | 65.8 (10.6)
Gender [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 12 | 14 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Difference in Visual-analog Score (VAS) for Anticipated Pain Prior to Injection and Actual Pain After Injection
Description: Members of both study groups completed the Visual Analog Scale (VAS) pain assessment both prior for anticipated pain and after injection for actual pain; these recorded scores were the primary study endpoint and were later compared to determine the difference in anticipated pain versus actual pain experienced. The VAS ranges from 0-10, where 0 is no pain and 10 is worst possible pain. The outcome measure is the mean anticipated pain minus the actual pain experienced.
Time Frame: Our outcome measure was collected within the 60 seconds before and following the steroid injection.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Triamcinolone (20 g) and 2% Lidocaine Injection Over A1 Pulley: Group one subjects received an injection of 0.5mL (20 g) of Triamcinolone and 0.5 mL of 2% Lidocaine over the A1 pulley.
  Triamcinolone (20 g) and 2% Lidocaine injection over the A1 pulley
  2% Lidocaine
  Triamcinolone (20 g)
- J-tip Lidocaine Administration, Then Steroid Injection: Group two subjects received a needle free "J-tip" administration of 0.5mL of 2% lidocaine prior (2-10 minutes) to needle injection of 0.5mL of Triamcinolone (20 g) over the A1 pulley.
  2% Lidocaine
  Triamcinolone (20 g)
  J-tip lidocaine administration
  Triamcinolone (20 g) Injection over the A1 pulley.
Arm/Group | Triamcinolone (20 g) and 2% Lidocaine Injection Over A1 Pulley | J-tip Lidocaine Administration, Then Steroid Injection
Number analyzed (Participants) | 29 | 31
units on a scale | 1.6 (0.44) | 2.8 (0.39)

ADVERSE EVENTS:
Arm/Group | Triamcinolone (20 g) and 2% Lidocaine Injection Over A1 Pulley | J-tip Lidocaine Administration, Then Steroid Injection
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No